CLINICAL TRIAL: NCT02442401
Title: Role of Negative Pressure Wound Therapy in Latissimus Dorsi Flap Donor Site Seroma Prevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Thana Laopiyasakul (Unknown); Pornthep Pungrasmi (Unknown); Poonpissamai Suwajo (Unknown)
Responsible Party: Principal Investigator, Apichai Angspatt, Apichai Angspatt, Chulalongkorn University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 030/55
Record Dates: First submitted 2015-05-10; First posted 2015-05-13 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: NPWT; Latissimus Dorsi Flap; Breast Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NPWT group (Experimental): Negative pressure wound therapy was used to prevent donor site seroma formation
  Interventions: Device: The negative pressure wound therapy
- Control group (No Intervention): Conventional method was used to the donor site

INTERVENTIONS:
Device: The negative pressure wound therapy
  Other Names: NPWT
  Arms: NPWT group

SUMMARY:
The use of NPWT as a post-operative dressing significantly reduces the incidence of seroma formation after harvesting LD flap.

DETAILED DESCRIPTION:
NPWT was left in place on donor site with constant pressure between -125 and -80 mmHg to reduce seroma formation

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-60 years Underwent breast reconstruction with LD Flap

Exclusion Criteria:

* Locally advanced cancer

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence of seroma | 3 months

SECONDARY OUTCOMES:
Aspirated Volume | 3 months
Frequency of Aspiration | 3 months